CLINICAL TRIAL: NCT01956825
Title: THE EFFECT OF DUAL TREATMENT WITH L-CARNITINE AND MAGNESIUM ON Patients With Non Alcoholic Fatty Liver Disease
Brief Title: The Effect Of Dual Treatment With L-Carnitine And Magnesium On Fatty Liver
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMC13023-13CTIL
Record Dates: First submitted 2013-09-12; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-09

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: non alcoholic fatty liver disease; LCARNITINE amino acid; magnesium; fat content
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water (Placebo Comparator): just water
- L-CARNITINE AND MAGNESIUM ("slim water" product) (Experimental): The experimental arm will receive a product "slim water", which contains 150 mg magnesium lactate and 2000 mg L-carnitine. The purpose is to follow the patients and examine several metabolic parameters over time (liver function test, lipid profile, liver fat content, etc.) and by that to show and prove the positive effect of the experimental treatment over placebo.
  Interventions: Dietary Supplement: "slim water"

INTERVENTIONS:
Dietary Supplement: "slim water"
  Arms: L-CARNITINE AND MAGNESIUM ("slim water" product)

SUMMARY:
The purpose of this study is to determine whether the dual therapy of the amino acid L-CARNITINE and magnesium have an effect on reducing the liver fat content in patients with non alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the dual therapy of the amino acid L-CARNITINE and magnesium have an effect on reducing the liver fat content in patients with non alcoholic fatty liver disease.

the study is an interventional one in which 60 patients who by definition have non alcoholic fatty licer disease (NAFLD) are divided randomly (double blind) into 2 groups: group 1: "study group". receive a product (flavoured water) which contains L-CARNITINE an magnesium. group 2: control. receive placebo. regular water. Length of trial - 12 weeks. The patients will be followed on a weekly base and variuos parameters will be compared (weight, lipid profile, insulin resistance etc.).

"fibrotest" will be used at the beginning of the trial and at the end (week 12) comparing the fat content before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

age>18, <80 y evidence to non alcoholic fatty liver disease

Exclusion Criteria:

age<18, >80 y pregnancy renal failure congestive heart failure active malignancy liver disease - etiology other than non alcoholic fatty liver disease (NAFLD). hypothyroidism/cushing total prenteral nutrition (TPN) in the last 6 month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
effect of LCARNITINE and magnesium treatment on the liver fat content | 12 weeks

SECONDARY OUTCOMES:
effect of L-CARNITINE and magnesium treatment on the metabolic panel | 12 weeks
  hepatic enzyme profile, lipid profile, weight, inflammatory markers, insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: DAN FELDMAN, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Hospital, Kfar Saba, Israel